CLINICAL TRIAL: NCT07334509
Title: Clinical Evaluation of a Simplified-Shade Nano-Hybrid Composite With Full-Coverage Silane Coating and High-Performance Pulverized Fillers Versus Conventional Multi-Shade Nano- Hybrid Composite in Direct Restoration of Posterior Proximal Carious Lesions After a 12- Month Follow-Up Period Using USPHS Criteria: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of a Simplified-Shade Nano-Hybrid Composite With Full-Coverage Silane Coating and High-Performance Pulverized Fillers
Acronym: FSC-HPC-GC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Raoh Kareem, Master's Degree Candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CONS-3-7-5
Record Dates: First submitted 2025-12-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Class II Dental Restorations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional multi shaded nano hybrid composite (Active Comparator): This group will receive the conventional multi shaded nano hybrid composite
  Interventions: Device: Conventional, multi shade nano, hybrid composite
- shaded nano hybrid composite (Experimental): Participants receive the simplified shaded nano hybrid composite restoration
  Interventions: Device: Simplified Nano hybrid composite

INTERVENTIONS:
Device: Simplified Nano hybrid composite — It's a simplified shade system for dental composite that is nano hybrid with full coverage saline coating and high performance pulverized fillers
  Arms: shaded nano hybrid composite
Device: Conventional, multi shade nano, hybrid composite — Traditional, multi shaded nano, hybrid, composite risen
  Arms: conventional multi shaded nano hybrid composite

SUMMARY:
The goal of this clinical trial is to evaluate simplified, shade, non-hybrid composite versus conventional multi Shade nano hybrid composite in class two restorations and reevaluate after one year follow up It's aim to answer Which composite has superior, anatomic form, color, match marginal, integrity, postoperative sensitivity, surface texture, and recurrent caries Researcher will compare the two composites And the participants will Have the restorations in posterior teeth and get a follow up after 12 months

ELIGIBILITY:
Inclusion Criteria:

* healthy human
* age ranging from18-64 years with a class two posterior restoration
* a fairly good oral hygiene
* teeth should be indicated for direct composite restoration
* teeth with vital pulp no symptoms of irreversible pulpitis
* patient who are willing to follow up after 12 months
* patient who have signed the informed consent

Exclusion Criteria:

* people under 18 years old or over 64 years old
* people with disabilities
* people with bad oral hygiene
* patient with systematic disease that could be affecting oral health
* cavities reaching the pulp
* people with periodontal diseases
* patient with parafunctional habits such as bruxism
* patient who are allergic to the restoration
* patients who are unwilling to follow after 12 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Marginal adaptation assessed using modified USPHS criteria | At baseline after six months after 1 year
  Marginal adaptation of the restorations will be clinically evaluated using the Modified United States Public Health Service (USPHS) criteria by a calibrated examiner.
  The scoring system includes the following categories:
  * Alpha (Score = 1): Excellent marginal adaptation, no visible gap
  * Bravo (Score = 2): Clinically acceptable marginal discrepancy
  * Charlie (Score = 3): Clinically unacceptable marginal defect requiring replacement
  The minimum score is 1 (best outcome) and the maximum score is 3 (worst outcome).
  Lower scores indicate better marginal adaptation, while higher scores indicate poorer marginal adaptation.